CLINICAL TRIAL: NCT01137864
Title: Impact of Infectious Diseases Specialists on the Appropriateness of Antimicrobial Therapy in Emergency Wards: a Multicenter Randomized Controlled Trial.
Brief Title: Impact of Infectious Diseases Specialists on the Appropriateness of Antimicrobial Therapy in Emergency Wards
Acronym: ATBREFEMERG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henri Mondor University Hospital (Other)
Responsible Party: Principal Investigator, Philippe LESPRIT, Dr Philippe LESPRIT, Henri Mondor University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREQHOS 08023b
Record Dates: First submitted 2010-06-01; First posted 2010-06-07 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Patients Under Antimicrobial Therapy
Keywords: Emergency wards; Hospitalization; Adults; Antimicrobial therapy
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infectious disease specialist advice (Experimental): Patients receiving the intervention (infectious disease specialist advice)
  Interventions: Other: Infectious disease specialist advice
- Control (No Intervention): Patients not receiving infectious disease specialist advice

INTERVENTIONS:
Other: Infectious disease specialist advice — Indication, choice, dosing and duration of antimicrobial therapy
  Arms: Infectious disease specialist advice

SUMMARY:
CONTEXT: Antibiotics are frequently used in hospital but the appropriateness of prescriptions ranged between 25-50%. The intervention of infectious disease specialists (IDS) could improve the appropriateness of prescriptions and reduce their use. The impact of IDS has not been yet fully estimated using a randomized trial to compare the quality of care of patients who will benefit of the intervention.

OBJECTIVES: To show using a randomized trial that patients hospitalized in emergency wards with IDS advice will receive more appropriate antimicrobial therapy but less exposure to antibiotics, as compared to patients who will not receive IDS advice.

METHODS: Prospective randomized trial comparing antibiotic exposure and appropriateness of prescriptions in two groups of patients admitted in emergency wards:

Control group: antibiotic prescriptions will be initiated and managed by the attending physicians Intervention group: antibiotic prescriptions will be systematically evaluated by the IDS and changed if judged necessary by the attending physicians, following IDS' advice.

STUDY PROCESS: The study will took place in the emergency wards of 4 university hospitals. For each ward, the period of the study will be 2 x 4 weeks.Total duration of the study: 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults Hospitalized in emergency wards Receiving antimicrobial therapy for active infection or prolonged surgical prophylaxis Therapy prescribed by the attending ward physician

Exclusion Criteria:

* Patients receiving antimicrobial therapy not prescribed by the attending ward physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Appropriateness of antimicrobial therapy | Between days 1 and 3
  Appropriateness of antimicrobial therapy will be evaluated at the end of hospitalization in emergency ward (on average, between days 1 and 3).

SECONDARY OUTCOMES:
Clinical impact | Between days 1 and 3
  Length of hospitalization; clinical outcome: resolution of infection; in hospital mortality. These end points will be evaluated at the end of hospitalization in emergency ward (on average, between days 1 and 3).
Antibiotic exposure | 14 days
  Antibiotic exposure will be evaluated at the time of discharge from emergency ward (on average, between days 1 and 3) using the following parameters:
  number of days of therapy/numbers of days of hospitalization; defined daily doses of antibiotic/number of days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lesprit, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor University Hospital, Créteil, France